CLINICAL TRIAL: NCT03362658
Title: Novel MRI Biomarkers for Monitoring Disease Progression in ALS
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other); Western University, Canada (Other); McGill University (Other); University of Toronto (Other); University of British Columbia (Other); Laval University (Other); University of Miami (Other); University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: RES0027887
Record Dates: First submitted 2017-10-18; First posted 2017-12-05 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
Keywords: Magnetic Resonance Imaging; MRI; Biomarker
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients: ALS patients (as well as patients with other related disorders such PLS, PMA, and ALS-FTD) will be recruited from ALS clinics under the direction of neurologists who are participating in this study. ALS patients should meet research criteria for suspected, possible, probable, probable laboratory supported, or definite ALS.
- Controls: Healthy controls who are age and gender matched to patients.

SUMMARY:
Routine MRI is normal in motor neuron diseases such as ALS. However, advanced MRI techniques can provide an objective measure of degeneration (a "biomarker") by examining brain structure, wiring, chemistry, and function. We will develop and evaluate novel MRI techniques that could improve our understanding of ALS and provide a means to diagnose it sooner and monitor its progression. Importantly, we expect these techniques to improve how new drugs are tested, which may lead to the more rapid discovery of a treatment for ALS.

Each participant will have 3 MRI scans over a period of 8 months, along with neurological and cognitive evaluations. Study visits will take 2 - 3 hours. MRI is a safe technique that does not involve radiation.

DETAILED DESCRIPTION:
Current clinical measures of disease burden have suboptimal sensitivity to disease progression in ALS. A biomarker would play an essential role in the evaluation of novel therapeutics, leading to the realization of effective treatments faster. Magnetic resonance imaging (MRI) holds promise as a non-invasive source of biomarkers in ALS. In this study data is collected from a national imaging platform (the Canadian ALS Neuroimaging Consortium [CALSNIC]) using standardized MRI and clinical protocols.

CALSNIC was founded with the objective to validate MRI biomarkers on a standardized multi-centre platform. CALSNIC is a multidisciplinary group of scientists at 7 centres across Canada. The first CALSNIC study entitled "MRI Biomarkers in ALS" (CALSNIC-1) is ongoing and slated to finish recruitment in 2017.

This study ("Novel MRI Biomarkers for Monitoring Disease Progression in ALS", CALSNIC-2) is a new project that will evaluate novel MRI biomarkers using advanced imaging acquisition and processing methods. The specific aims of CALSNIC-2 are 1) to establish a standardized MRI and clinical protocol across the 7 centres, and 2) to validate MRI measures with clinical measures of disease burden and progression.

It is anticipated that the project will lead to the discovery of MR-based biomarkers of cerebral degeneration that can be applied across different centres and hence, can assist with drug development. Secondly, this project will expand CALSNIC to include more centres and provide opportunities for collaborative and multidisciplinary translational research on a national scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a suspected or confirmed diagnosis as described in Study Populations
* For those with a diagnosis of ALS, patients will be considered with an El Escorial classification of suspected, possible, probable, probable lab-supported, and definite ALS.
* Patients 18 years of age or older
* Healthy controls over the age of 40.
* Be able to lie in an MRI machine for approximately 60 minutes

Exclusion Criteria:

* Subjects with psychiatric/CNS illnesses such as Major Depressive Disorder, Schizophrenia, and Bipolar disorder.
* Subjects with significant head injury or other neurological disease (stroke, brain tumour).
* Subjects ineligible for MRI investigation due to a pacemaker or other metallic foreign body.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients with a diagnosis of motor neuron disease (MND). This includes the diagnoses of amyotrophic lateral sclerosis (ALS), primary lateral sclerosis (PLS), and progressive muscular atrophy (PMA).
  2. Patients with frontotemporal dementia (FTD) with or without motor neuron signs.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-10; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cortical thickness in millimetres. | 8 months
  This primary analysis will evaluate neuronal integrity at baseline and specified follow up periods. Patients and controls scans will be compared.
Change in DTI indices (unitless). | 8 months
  This primary analysis will evaluate white matter integrity at baseline and specified follow up periods. Patients and controls scans will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kalra, MD, Principal Investigator — FRCPC
Locations (9):
- United States (2):
  - University of Miami, Miami, Florida
  - University of Utah, Salt Lake City, Utah
- Canada (7):
  - University of Calgary / Heritage Medical Research Clinic, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia / GF Strong Rehab Centre, Vancouver, British Columbia
  - Western University / London Health Sciences Centre, London, Ontario
  - University of Toronto / Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University / Montreal Neurological Institute and Hospital, Montreal, Quebec
  - Laval University, Québec, Quebec